CLINICAL TRIAL: NCT06839378
Title: Fluorouracil-labeled Nascent RNA Technology for Evaluating the Effects of Different Hyperthermic Intraperitoneal Chemotherapy Regimens on the Transcriptome of Pseudomyxoma Peritonei
Brief Title: Flura-seq for Evaluating the Effects of Different Hyperthermic Intraperitoneal Chemotherapy Regimens on the Transcriptome of Pseudomyxoma Peritonei
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tsinghua Chang Gung Hospital (Other)
Collaborators: Tsinghua University (Other)
Responsible Party: Principal Investigator, Yan Li, Director of Department of Surgical Oncology, Beijing Tsinghua Chang Gung Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 24753-0-02
Record Dates: First submitted 2025-02-17; First posted 2025-02-21 (Actual); Results first posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Pseudomyxoma Peritonei
Keywords: Flura-seq; PMP; HIPEC; Fluorouracil-labeled Nascent RNA Technology
MeSH Terms: conditions — Pseudomyxoma Peritonei | interventions — Fluorouracil

STUDY DESIGN:
Intervention Model Description: This study is a single-center, double-arm, open-label exploratory clinical study. The patients will be randomly divided into cisplatin group and cisplatin + docetaxel group, each group contains 18 patients. 5-FU (400 mg/m2) will be injected IV bolus before operation. After CRS, the patients will be treated with cisplatin or cisplatin + docetaxel HIPEC respectively. The tumor tissue samples of patients will be collected before and after HIPEC treatment. The tumor tissue samples before and after HIPEC treatment will be sequenced by Flura-seq using high-throughput sequencing technology, and the changes of newly generated transcripts in tumor tissue during HIPEC will be analyzed. The differentially expressed genes in the cisplatin group and the cisplatin + docetaxel group will be compared to evaluate the effect of different HIPEC regimens on the transient transcriptome of PMP tumor. It lays a foundation for optimizing HIPEC regimen and judging new therapeutic targets.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cisplatin Group (Experimental): After completing CRS, the patient will undergo cisplatin HIPEC treatment. Add 120 mg of cisplatin to 3000 ml of physiological saline, heat to 43 ℃, perfuse at a flow rate of 400 ml/min, and perfuse for 60 minutes.
  Interventions: Procedure: intravenously inject with 5-FU (400 mg/m2)
- Cisplatin + Docetaxel Group (Active Comparator): After completing CRS, the patient will undergo HIPEC treatment with cisplatin and docetaxel. Add 120 mg of docetaxel and 120 mg of cisplatin to 3000 ml of physiological saline, heat to 43 ℃, perfuse at a flow rate of 400 ml/min, and perfuse for 60 minutes.
  Interventions: Procedure: intravenously inject with 5-FU (400 mg/m2)

INTERVENTIONS:
Procedure: intravenously inject with 5-FU (400 mg/m2) — 5-FU (400 mg/m2) will be injected IV bolus before operation. After CRS, the patients will be treated with cisplatin or cisplatin + docetaxel HIPEC respectively. The tumor tissue samples of patients will be collected before and after HIPEC treatment. The tumor tissue samples before and after HIPEC treatment will be sequenced by Flura-seq using high-throughput sequencing technology, and the changes of newly generated transcripts in tumor tissue during HIPEC will be analyzed. The differentially expressed genes in the cisplatin group and the cisplatin + docetaxel group will be compared to evaluate the effect of different HIPEC regimens on the transient transcriptome of PMP tumor.

SUMMARY:
The main objective of this study is to combine HIPEC regimens with Flura-seq to detect the effects of different HIPEC regimens (cisplatin vs. cisplatin+ docetaxel) on the nascent transcriptome of PMP tumors, so as to quantitatively assess the efficacy of different HIPEC regimens in the early stage, and to lay the foundation for optimizing the HIPEC regimens and exploring new therapeutic targets.

DETAILED DESCRIPTION:
1. Participants:

   ① Diagnosed PMP patients;

   ② Patients can receive CRS+HIPEC treatment.
2. Trial protocol: the patients will be randomly divided into cisplatin group and cisplatin + docetaxel group. Preoperative intravenous bolus injection of 5-FU (400 mg/m2) will be given before CRS+HIPEC treatment. After CRS, the patients will be treated with cisplatin or cisplatin + docetaxel HIPEC, respectively. Cisplatin 120 mg or docetaxel 120 mg + Cisplatin 120 mg will be added to 3,000 ml of saline, heated to 43 ℃, and perfused at a flow rate of 400 ml/min for 60 min.
3. Sample collection: tumor tissue samples (5-10 g) will be collected before and after HIPEC treatment, and will be stored at 80 ℃ for nascent transcriptome sequencing.
4. Sequencing analysis of nascent transcriptome: using high-throughput sequencing technology, the RNA extracted from tumor tissue samples before and after treatment with cisplatin or cisplatin + docetaxel HIPEC will be sequenced by Flura-seq to analyze the changes of newly synthesized transcripts in tumor tissue during HIPEC.
5. Data analysis: the sequencing data will be processed and analyzed by bioinformatics methods. The differentially expressed genes in cisplatin group and cisplatin + docetaxel group will be compared to evaluate the efficacy of different HIPEC regimens on PMP. Functional annotation and pathway analysis of differentially expressed genes will be performed to explore molecular therapeutic targets for PMP-specific RNA.
6. Treatment regimen for poor therapeutic effect: the study will not change the patient's existing HIPEC regimen. If the results show that HIPEC is not effective in treating the patient, it means that the drug is not effective for the patient during subsequent chemotherapy, and the chemotherapy regimen can be adjusted accordingly based on the Flura-seq results.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years old, regardless of gender and race;
* Pathologically confirmed as pseudomyxoma peritonei; acceptable for CRS+HIPEC treatment;
* KPS score ≥ 60, with expected survival time more than 12 months;
* The functions of important organs are basically normal, with no significant abnormalities in liver or kidney function;
* No history of allergy to biological products;
* No serious bacterial or viral infection;
* Non-pregnancy and lactation;
* The patient or his/her delegate understands and cooperates with the treatment and signs the informed consent for the treatment.

Exclusion Criteria:

* Highly allergic or with a history of severe allergies, especially to biological products;
* Shock, systemic failure, unstable vital signs, and inability to cooperate with the examination;
* Those who have mental or psychological diseases and cannot cooperate with treatment and curative effect evaluation;
* T-lymphocyte carcinoma/tumor;
* Patients with systemic infection or severe local infection requiring anti-infection treatment;
* Complicated with dysfunction of heart, lung, brain, kidney, liver and other important organs;
* Coagulation disorders (e.g., hemophilia);
* Infectious diseases (e.g. HIV, RPR, active TB, etc.);
* Pregnant or lactating women, or women who have pregnancy plans within half a year;
* Patients who are taking immunosuppressive drugs or long-term anti-rejection drugs after organ transplantation;
* Patients with severe autoimmune diseases;
* Any life-threatening disease, physical condition or organ system dysfunction that the researcher believes may damage the safety of subjects and expose the research results to unnecessary risks; Drug-dependent persons;
* Patients and/or authorized family members who refuse or do not actively sign the informed consent;
* Participants in other clinical studies within 3 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2025-02-17 (Actual); Primary Completion 2025-08-06 (Actual); Study Completion 2025-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yan Li, PhD, Principal Investigator — Beijing Tsinghua Changgeng Hospital
Locations (1):
- Beijing Tsinghua Changgung Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
Sequencing raw data
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: From 2025 to 2028
Access Criteria: For information sharing, contact the PI to access the IPD

REFERENCES:
- [Background] Wang Q, Lu F, Lan R. RNA-sequencing dissects the transcriptome of polyploid cancer cells that are resistant to combined treatments of cisplatin with paclitaxel and docetaxel. Mol Biosyst. 2017 Sep 26;13(10):2125-2134. doi: 10.1039/c7mb00334j. PMID 28825433
- [Background] Mehta AM, Huitema AD, Burger JW, Brandt-Kerkhof AR, van den Heuvel SF, Verwaal VJ. Standard Clinical Protocol for Bidirectional Hyperthermic Intraperitoneal Chemotherapy (HIPEC): Systemic Leucovorin, 5-Fluorouracil, and Heated Intraperitoneal Oxaliplatin in a Chloride-Containing Carrier Solution. Ann Surg Oncol. 2017 Apr;24(4):990-997. doi: 10.1245/s10434-016-5665-6. Epub 2016 Nov 28. PMID 27896510
- [Background] Basnet H, Tian L, Ganesh K, Huang YH, Macalinao DG, Brogi E, Finley LW, Massague J. Flura-seq identifies organ-specific metabolic adaptations during early metastatic colonization. Elife. 2019 Mar 26;8:e43627. doi: 10.7554/eLife.43627. PMID 30912515
- [Background] Fernandez RN, Daly JM. Pseudomyxoma peritonei. Arch Surg. 1980 Apr;115(4):409-14. doi: 10.1001/archsurg.1980.01380040037006. PMID 7362446
- [Background] Chua TC, Moran BJ, Sugarbaker PH, Levine EA, Glehen O, Gilly FN, Baratti D, Deraco M, Elias D, Sardi A, Liauw W, Yan TD, Barrios P, Gomez Portilla A, de Hingh IH, Ceelen WP, Pelz JO, Piso P, Gonzalez-Moreno S, Van Der Speeten K, Morris DL. Early- and long-term outcome data of patients with pseudomyxoma peritonei from appendiceal origin treated by a strategy of cytoreductive surgery and hyperthermic intraperitoneal chemotherapy. J Clin Oncol. 2012 Jul 10;30(20):2449-56. doi: 10.1200/JCO.2011.39.7166. Epub 2012 May 21. PMID 22614976
- [Background] Hinson FL, Ambrose NS. Pseudomyxoma peritonei. Br J Surg. 1998 Oct;85(10):1332-9. doi: 10.1046/j.1365-2168.1998.00882.x. PMID 9782010
- [Background] Carr NJ, Cecil TD, Mohamed F, Sobin LH, Sugarbaker PH, Gonzalez-Moreno S, Taflampas P, Chapman S, Moran BJ; Peritoneal Surface Oncology Group International. A Consensus for Classification and Pathologic Reporting of Pseudomyxoma Peritonei and Associated Appendiceal Neoplasia: The Results of the Peritoneal Surface Oncology Group International (PSOGI) Modified Delphi Process. Am J Surg Pathol. 2016 Jan;40(1):14-26. doi: 10.1097/PAS.0000000000000535. PMID 26492181
- [Background] Ramaswamy V. Pathology of Mucinous Appendiceal Tumors and Pseudomyxoma Peritonei. Indian J Surg Oncol. 2016 Jun;7(2):258-67. doi: 10.1007/s13193-016-0516-2. Epub 2016 Mar 19. PMID 27065718
- [Background] Smeenk RM, Bruin SC, van Velthuysen ML, Verwaal VJ. Pseudomyxoma peritonei. Curr Probl Surg. 2008 Aug;45(8):527-75. doi: 10.1067/j.cpsurg.2008.04.003. No abstract available. PMID 18590843

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was conducted at a single-center hospital (Beijing Tsinghua Changgung Hospital, Department of Peritoneal Oncology) from February 17, 2025, to August 6, 2025. Potential participants were identified through outpatient clinics and physician referrals. All screened individuals underwent preliminary eligibility assessment based on the study's inclusion and exclusion criteria.
Pre-assignment Details: After providing informed consent, 36 enrolled participants entered a screening phase to confirm eligibility based on predefined inclusion/exclusion criteria. All 36 participants successfully completed screening and proceeded to randomization. No participants were excluded or withdrew during this phase. Using a randomization table provided by the Beijing Tsinghua Changgung Hospital Clinical Data Management Center, the 36 participants were randomly assigned to two groups (18 participants per group
Groups:
- Experimental : Cisplatin Group; Active Comparator : Cisplatin + Docetaxel Group: 5-FU (400 mg/m²) has been injected IV bolus before operation. After CRS, the patients have been treated with cisplatin or cisplatin + docetaxel HIPEC respectively. The tumor tissue samples of patients have been collected before and after HIPEC treatment. The tumor tissue samples before and after HIPEC treatment have been sequenced by Flura-seq using high-throughput sequencing technology, and the changes of newly generated transcripts in tumor tissue during HIPEC have been analyzed. The differentially expressed genes in the cisplatin group and the cisplatin + docetaxel group have been compared to evaluate the effect of different HIPEC regimens on the transient transcriptome of PMP tumor.
Period: Overall Study
Arm/Group | Experimental : Cisplatin Group | Active Comparator : Cisplatin + Docetaxel Group
Started | 18 | 18
Completed | 18 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All 36 participants who were randomized and assigned to the two study arms (18 per group) are included in the baseline analysis. There was no discrepancy between the number of participants enrolled, randomized, and included in the baseline characteristics analysis. No participants were excluded post-randomization prior to baseline assessment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental : Cisplatin Group | Active Comparator : Cisplatin + Docetaxel Group | Total
Number analyzed (Participants) | 18 | 18 | 36
Age, Customized [Count of Participants; unit: Participants] — Age 18-75 years old, regardless of gender and race
  Participants
    Age 18-75 years old | 18 | 18 | 36
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 19
  Male | 9 | 8 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 18 | 18 | 36
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 18 | 18 | 36
  Unknown or Not Reported | 0 | 0 | 0
Histological characteristics of 36 PMP patients treated with CRS+HIPEC [Count of Participants; unit: Participants] — The four level classification (Acellular mucus, low-grade mucinous carcinoma peritoneum, high-grade mucinous carcinoma peritoneum, high-grade mucinous carcinoma peritoneum with signet ring cells) is based on the 2016 Peritoneal Surface Oncology Group International (PSOGI) consensus classification standard.
  Participants
    Acellular mucus | 0 | 1 | 1
    low-grade mucinous carcinoma peritoneum | 10 | 12 | 22
    high-grade mucinous carcinoma peritoneum | 5 | 5 | 10
    high-grade mucinous carcinoma peritoneum with sign | 3 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Changes in RNA in Tumor Tissues Before and After HIPEC
Description: Main index parameters: information on the amount of differentially expressed genes and the magnitude of change between the cisplatin group and the cisplatin+ docetaxel group. The amount of differentially expressed genes is expressed as mean ± standard deviation and statistically analyzed by t-test or rank-sum test, and the comparison between groups is performed by unpaired t-test. Differences are considered statistically significant when P< 0.05. Based on the statistical results, the efficacy of the two HIPEC regimens (cisplatin or cisplatin+ docetaxel) on PMP will be analyzed.
  Expected results and clinical interpretation: More changes in newly generated RNA in the tumor tissue indicate a greater impact of HIPEC on the transcriptome of the tumor cells, possibly indicating better efficacy.
Time Frame: From the initiation of Cytoreductive Surgery (CRS) to the completion of Hyperthermic Intraperitoneal Chemotherapy (HIPEC). CRS takes 4-8 hours, HIPEC takes 1 hour. Pre and post-HIPEC tumor tissues were collected for RNA-sequencing.
Measure: Mean (Standard Deviation); unit: Numbers of changed RNA
Arm/Group | Experimental : Cisplatin Group | Active Comparator : Cisplatin + Docetaxel Group
Number analyzed (Participants) | 18 | 18
Numbers of changed RNA | 1413 (876) | 1927 (992)

2. Secondary Outcome: Comparison of Transcriptomic Changes Detected by Flura-seq vs. Bulk RNA-seq
Description: This secondary outcome quantifies and compares differentially expressed genes (DEGs) identified via Flura-seq (spatial transcriptomics) and bulk RNA-seq methodologies across all samples collected before and after hyperthermic intraperitoneal chemotherapy (HIPEC).
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: Numbers of changed RNA
Groups:
- Transcriptomic Changes Detected by Flura-seq: This secondary outcome quantifies and compares differentially expressed genes (DEGs) identified via Flura-seq (spatial transcriptomics) methodologies across all samples collected before and after hyperthermic intraperitoneal chemotherapy (HIPEC).
- Transcriptomic Changes Detected by Bulk RNA-seq: This secondary outcome quantifies differentially expressed genes (DEGs) identified via bulk RNA-seq methodologies across all samples collected before and after hyperthermic intraperitoneal chemotherapy (HIPEC).
Arm/Group | Transcriptomic Changes Detected by Flura-seq | Transcriptomic Changes Detected by Bulk RNA-seq
Number analyzed (Participants) | 36 | 36
Numbers of changed RNA | 1,690 (940) | 340 (300)

ADVERSE EVENTS:
Time Frame: From the end of CRS+HIPEC treatment to 30 days after surgery.
Description: The analysis population comprised all 36 enrolled patients who met the pre-specified inclusion and exclusion criteria. This clinical trial mainly collected Grade 3 - 4 serious adverse events. Other non-serious adverse events are not systematically collected or reported.
Arm/Group | Cisplatin Group | Cisplatin + Docetaxel Group
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cisplatin Group (N=18) | Cisplatin + Docetaxel Group (N=18)
Venous Thromboembolism Occurrence (time, symptoms and signs, ultrasound/CTA, measures, prognosis) (General disorders) | 0 | 0 — Details on time, symptoms, diagnostic imaging (ultrasound/CTA), treatment measures and prognosis. May be related to surgical intervention. Assessed through clinical records.
Symptomatic Deep - Vein Thrombosis (General disorders) | 0 | 0 — Detected by clinical symptoms, signs and confirmed via ultrasound. Associated with post - operative or high - risk conditions.
Pulmonary Embolism (Vascular disorders) | 0 | 0 — Diagnosed by CTA. Symptoms include dyspnea, chest pain. Can be life - threatening and related to VTE risk factors.
Post - operative Gastrointestinal Fistula (Gastrointestinal disorders) | 0 | 0 — Identified through clinical examination and imaging techniques.
Bone Marrow Suppression (Blood and lymphatic system disorders) | 0 | 0 — Assessed by blood cell counts (WBC, RBC, platelets). Graded according to severity.
Intestinal Obstruction (Gastrointestinal disorders) | 0 | 0 — Symptoms are abdominal pain, vomiting, constipation. Diagnosed by clinical presentation and imaging.
Urinary Tract Infection (Renal and urinary disorders) | 0 | 0 — Diagnosed by urine tests and symptoms like frequency, urgency. Treated with antibiotics.
Urinary Fistula (Renal and urinary disorders) | 0 | 0 — Detected by abnormal urine leakage, imaging is used for further evaluation.
Renal Insufficiency (Renal and urinary disorders) | 0 | 0 — Assessed by serum creatinine, BUN, eGFR. Severe cases may need dialysis.
Massive Hemorrhage (Blood and lymphatic system disorders) | 0 | 0 — Defined by significant blood loss and low hemoglobin levels. May require blood transfusion.
Respiratory system (pneumonia, pleural effusion, pneumothorax) (Respiratory, thoracic and mediastinal disorders) | 0 | 0 — Diagnosed by clinical symptoms and chest imaging.
Circulatory system (arrhythmia, hypotension, ischemic cardiomyopathy, pulmonary edema) (Cardiac disorders) | 0 | 0 — Assessed by ECG, blood pressure monitoring, imaging. May be related to anesthesia or post - op state.
Nervous system (stroke, neurological paralysis) (Nervous system disorders) | 0 | 0 — Diagnosed by neurological examination and brain imaging.
Intra - abdominal Infection (Infections and infestations) | 0 | 0 — Detected by abdominal pain, fever, and imaging showing fluid collection.
Incision dehiscence, infection (Skin and subcutaneous tissue disorders) | 0 | 0 — Visually inspected for dehiscence, swabbed for infection testing.
Venous catheterization (septicemia, embolism, pneumothorax) (Injury, poisoning and procedural complications) | 0 | 0 — Detected by clinical symptoms and imaging.

LIMITATIONS AND CAVEATS:
The case number is limited as PMP is a rare disease. Conducting future multicenter studies could potentially facilitate the accumulation of a larger sample size, thereby enabling more robust analyses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-11-01): https://cdn.clinicaltrials.gov/large-docs/78/NCT06839378/Prot_SAP_000.pdf